CLINICAL TRIAL: NCT03699995
Title: Imaging Modalities for Melanoma Screening and Diagnosis
Brief Title: MoleMapper, Visiomed, and Confocal Microscopy in Screening Participants for Melanoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Sancy A Leachman, MD, PhD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY00018408; NCI-2018-01152 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018408 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Melanoma; Melanocytic Nevus; Skin Carcinoma
MeSH Terms: conditions — Melanoma; Nevus, Pigmented | interventions — Microscopy, Confocal; Dermoscopy; X-Rays; Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (imaging, biopsy) (Experimental): Participants undergo imaging of suspicious moles via smartphone app MoleMapper/Sklip app/native smartphone camera app, digital dermoscopy, and confocal microscopy. Participants then receive lidocaine SC and undergo shave or punch biopsy of suspected melanomas.
  Interventions: Other: Confocal Microscopy; Other: Dermoscopy; Procedure: Imaging Procedure; Drug: Lidocaine; Procedure: Punch Biopsy; Procedure: Shave Biopsy

INTERVENTIONS:
Other: Confocal Microscopy — Undergo confocal microscopy
  Other Names: Confocal Laser Scanning Microscopy
Other: Dermoscopy — Undergo digital dermoscopy
Procedure: Imaging Procedure — Undergo MoleMapper/Sklip app/native smartphone camera app imaging with smartphone
  Other Names: Diagnostic Imaging Technique; Imaging; Imaging Procedures; Imaging Technique; imaging type; imaging_type; Medical Imaging
Drug: Lidocaine — Given SC
  Other Names: .omega.-Diethylamino-2,6-dimethylacetanilide; 2-(Diethylamino)-2',6'-acetoxylidide; Cuivasil; Duncaine; Leostesin; Lidothesin; Lignocaine; Rucaina
Procedure: Punch Biopsy — Undergo punch biopsy
  Other Names: Punch Biopsy of Skin
Procedure: Shave Biopsy — Undergo shave biopsy

SUMMARY:
This trial studies how well MoleMapper, Visiomed, and confocal microscopy work in screening participants for melanoma. Analyzing images (photographs) made with three different portable imaging systems may be as good as a visit to a dermatologist's office for finding melanomas before they can spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the clinical utility of clinical images, digital dermoscopy images and in-vivo confocal microscopy for teledermatology.

SECONDARY OBJECTIVE:

I. To incorporate in vivo confocal images into the triage system in order to determine to what degree the information gathered in this modality changes the classification of a lesion assigned by a licensed dermatologist.

TERTIARY OBJECTIVE:

I. To assess the potential improvement of virtual patient triage when adding digital dermoscopy images to clinical images presented by patients to their provider (via e-visit or e-consult).

OUTLINE:

Participants undergo imaging of suspicious moles via smartphone application (app) MoleMapper/Sklip app/native smartphone camera app, digital dermoscopy, and confocal microscopy. Participants then receive lidocaine subcutaneously (SC) and undergo shave or punch biopsy of suspected melanomas.

After completion of study intervention, patients are followed up within 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Persons who participate in the free skin cancer screening at the PDX Skincare Festival at Oregon Health & Science University (OHSU) in 2021/2022 (date pending) and are informed by a provider that they have a pigmented lesion for which a biopsy is recommended are potentially eligible to participate in this study.
* Persons who participate in the free skin cancer screening at the War on Skin Cancer event at OHSU in 2021/2022 (date pending) or other dates and locations and are informed by a provider that they have a clinically benign or atypical nevi are eligible to participate in the imaging portion of this study. No biopsy will be offered to these participants.
* Persons age 18-80 are eligible for the study
* Persons of any sex can be enrolled.
* Persons of any race are eligible but we anticipate that most participants will be Non-Hispanic whites due to the prevalence of melanoma and other skin cancers in this group.
* Only persons who can provide signed statement of informed consent will be enrolled.
* Persons who are identified in OHSU Dermatology clinics or through OHSU e-visit and e-consult platforms as having a skin lesion in need of a biopsy for skin cancer
* Persons identified via the Melanoma Community Registry (MCR) (IRB approved: 00010561)

Exclusion Criteria:

* Allergy to the anesthetic (lidocaine).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the imaging modalities | Up to 1 year
  Sensitivity is defined as recommend immediate biopsy (red) lesions correctly identified as red by the dermatologists. The nature of statistical data analyses will be descriptive and exploratory to estimate effect sizes and their variation as well as generate hypotheses for the future study design. Sensitivity and specificity will be estimated along with exact 95% confidence intervals.
Specificity of imaging modalities | Up to 1 year
  Specificity is defined as green (follow-up at annual skin exam) or yellow lesions (recommend examination by dermatologist in 3 months) correctly identified. The nature of statistical data analyses will be descriptive and exploratory to estimate effect sizes and their variation as well as generate hypotheses for the future study design. Sensitivity and specificity will be estimated along with exact 95% confidence intervals.

SECONDARY OUTCOMES:
Sensitivity by changes after consideration of in vivo reflectance mode confocal scanning laser microscopy (RCM) report | Up to 1 year
  Secondary analysis will be done with the biopsied lesions that were analyzed by RCM. The dermatologists will be provided a report of the RCM findings as well as the VisioMed images and asked to make the same classification as above. Changes in sensitivity and specificity will be determined.
Specificity by changes after consideration of RCM report | Up to 1 year
  Secondary analysis will be done with the biopsied lesions that were analyzed by RCM. The dermatologists will be provided a report of the RCM findings as well as the Visiomed images and asked to make the same classification as above. Changes in sensitivity and specificity will be determined.

OTHER OUTCOMES:
Improvements in virtual triage of patients when enabling patients to take and submit digital dermoscopy images from home | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Ludzik, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Sancy Leachman, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided